CLINICAL TRIAL: NCT05684471
Title: Comparison of the Efficiency of Ultrasound-Guided Suprainguinal Fascia Iliaca Block and Anterior Quadratus Lumborum Block in Patients Undergoing Total Hip Arthroplasty Under Spinal Anesthesia
Brief Title: SFIB vs Anterior QLB in Total Hip Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsun University (Other)
Responsible Party: Principal Investigator, Serkan Tulgar, Principal Investigator, Samsun University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LINRA
Record Dates: First submitted 2023-01-05; First posted 2023-01-13 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Pain
Keywords: Postoperative pain management; Total hip arthroplasty; Suprainguinal fascia iliaca block; Anterior QLB
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound Guided Suprainguinal Fascia iliaca Block (Active Comparator): Patients randomized to receive suprainguinal fascia iliaca block
  Interventions: Procedure: Ultrasound Guided Suprainguinal Fascia iliaca Block
- Ultrasound Guided Anterior quadratus lumborum block (Active Comparator): Patients randomized to receive anterior quadratus lumborum block
  Interventions: Procedure: Ultrasound Guided Anterior Quadratus Lumborum Block

INTERVENTIONS:
Procedure: Ultrasound Guided Suprainguinal Fascia iliaca Block — Patients in this group will be administered SFIB with 50 mL of local anesthetic solution (Bupivacaine %0.25) under ultrasound guidance after the surgery is completed.
  Arms: Ultrasound Guided Suprainguinal Fascia iliaca Block
Procedure: Ultrasound Guided Anterior Quadratus Lumborum Block — Patients in this group will be administered anterior QLB with 40 mL of local anesthetic (Bupivacaine %0.25) under ultrasound guidance after the surgery is completed.
  Arms: Ultrasound Guided Anterior quadratus lumborum block

SUMMARY:
Quadratus lumborum block (QLB) is a facial plane block defined to provide analgesia from T7-L3 dermatomes. There are articles reporting that it is an effective analgesic method in hip surgeries. Suprainguinal fascia iliaca block (SIFIB) also blocks components of the lumbar plexus and provides effective analgesia in hip surgeries. The investigators aim to compare the effectiveness of QLB and SIFIB in patients undergoing primary total hip arthroplasty (THA).

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) classification I-II-III
* Scheduled for total hip artroplasty surgery under spinal anesthesia

Exclusion Criteria:

* Patients who did not want to participate in the study
* Patients with cognitive dysfunction who cannot evaluate the NRS score and cannot use PCA
* Known local anesthetics and opioid allergy,
* Pregnancy or lactation
* Patients with a contraindication to spinal and regional anesthesia
* Presence of multiple fractures

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2023-01-18 (Actual); Primary Completion 2024-05-07 (Actual); Study Completion 2024-05-07 (Actual)

PRIMARY OUTCOMES:
Cumulative opioid comsumption | up to 24 hour
  Morphine consumptions for both group will be recorded

SECONDARY OUTCOMES:
Numeric rating scale for postoperative pain intensity | up to 24 hours
  Changes in Numeric Rating Scale (NRS) at rest and on movement will be recorded at intervals. (3-6-12-18-24th hour) NRS is a unidimensional measure of pain intensity in adults. The NRS is a segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of his/her pain. The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable").
Quality of Recovery (QoR-15) | at 24th hour
  The impact of surgical and anesthetic interventions on perioperative quality of life and ability to resume routine life activities will be assessed using the Quality of Recovery (QoR) tool. The QoR-15 scale is a patient-based outcome measure in the form of a 15-item validated questionnaire.
Presence of quadriceps motor block (defined as paralysis or paresis). | up to 24 hours
  Quadriceps motor function will be tested with the patient supine and with the hip and knee flexed at 45º and 90º, respectively. The subject will be asked to extend the knee first against gravity and then against resistance. Quadriceps strength will be graded according to a 3-point scale: normal strength = 0 point (extension against resistance); paresis = 1 point (extension against gravity but not against resistance); and paralysis = 2 points (no extension).

CONTACTS AND LOCATIONS:
Overall Officials: Serkan Tulgar, Principal Investigator — Samsun Üniversitesi tıp fakültesi, Samsun Eğitim ve Araştırma Hastanesi
Locations (1):
- Samsun University, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] James M, Bentley RA, Womack J, Goodman BA. Safety profile and outcome after ultrasound-guided suprainguinal fascia iliaca catheters for hip fracture: a single-centre propensity-matched historical cohort study. Can J Anaesth. 2022 Sep;69(9):1139-1150. doi: 10.1007/s12630-022-02279-0. Epub 2022 Jul 12. PMID 35819630
- [Background] Wang Q, Hu J, Zhang W, Zeng Y, Yang J, Kang P. Comparison Between Ultrasound-Guided Suprainguinal Fascia Iliaca Block and Anterior Quadratus Lumborum Block for Total Hip Arthroplasty: A Prospective, Double-Blind, Randomized Controlled Trial. J Arthroplasty. 2022 Apr;37(4):763-769. doi: 10.1016/j.arth.2022.01.011. Epub 2022 Jan 11. PMID 35026362
- [Background] Shamim R, Prasad G, Bais PS, Priya V, Singh TK, Ambasta S, Philips AK. Ultrasound-Guided Suprainguinal Fascia Iliaca Compartment Block for Postoperative Analgesia in Patients Undergoing Hip and Femur Surgeries: A Retrospective Analysis. Anesth Essays Res. 2020 Jul-Sep;14(3):525-530. doi: 10.4103/aer.AER_9_21. Epub 2021 Mar 22. PMID 34092870